CLINICAL TRIAL: NCT03700541
Title: Influence of Peri-operative Opioid Analgesia on Circulating Tumor Cells in Patients Undergoing Laparoscopic Colorectal Cancer Surgery - Multi-center, Randomized Clinical Trial
Brief Title: Influence of Opioid Analgesia on Circulating Tumor Cells in Laparoscopic Colorectal Cancer Surgery
Acronym: POACC-2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Institute of Molecular and Translational Medicine, Czech Republic (Other)
Collaborators: General University Hospital, Prague (Other); Tomas Bata Hospital, Czech Republic (Other); University Hospital Ostrava (Other); Hospital Novy Jicin (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: POACC-2
Record Dates: First submitted 2018-10-03; First posted 2018-10-09 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-09

CONDITIONS: Colorectal Cancer; Circulating Tumor Cell
Keywords: Perioperative analgesia; Colorectal Cancer; Circulating Tumor Cell
MeSH Terms: conditions — Colorectal Neoplasms; Neoplastic Cells, Circulating | interventions — Morphine; Pirinitramide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Morphine (Active Comparator): Morphine-based perioperative analgesia
  Interventions: Drug: Morphine
- Piritramid (Active Comparator): Piritramid-based perioperative analgesia
  Interventions: Drug: Piritramid

INTERVENTIONS:
Drug: Morphine — Morphine intravenous
  Arms: Morphine
Drug: Piritramid — Piritramid intravenous
  Arms: Piritramid

SUMMARY:
To compare the effects of three types of perioperative analgesia on the number of circulating tumor cells following radical colorectal cancer surgery. To find correlations with other perioperative factors and clinical/pathological disease characteristics.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing open radical surgery for colorectal cancer
* age over 18 years
* signed informed consent

Exclusion Criteria:

* intolerance of the study drugs
* history of CRC surgery
* neoadjuvant therapy
* other malignancy not in permanent remission
* chronic opioid medication or opioid administration within 7 days preoperatively
* immunosuppressive or corticosteroid therapy
* surgery within 30 days preoperatively (except minor)
* chronic or acute infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-12-06 (Actual)

PRIMARY OUTCOMES:
Change in number of circulating tumor cells prior to surgery to 2 - 4 weeks after surgery | 1 - 3 days before surgery to 4 weeks after surgery
  Baseline number of circulating tumor cells will be recorded prior to surgery in a venous blood sample. Number of circulating tumor cells will be measured 2 - 4 weeks after surgery in a venous blood sample. These two values will be compared.

SECONDARY OUTCOMES:
Pain assessment | Time Frame: 3 days postoperatively
  Pain intensity assessed using Numerical Rating Scale (0-10)

CONTACTS AND LOCATIONS:
Overall Officials: Marian Hajduch, MD PhD, Principal Investigator — Institute of Molecular and Translational Medicine, Palacky University, Olomouc
Locations (3):
- Czechia (3):
  - T. Bata Regional Hospital Zlin, Zlin, South Moravian
  - University Hospital Ostrava, Ostrava
  - General University Hospital, Prague

IPD SHARING:
Plan to Share IPD: No